CLINICAL TRIAL: NCT03162536
Title: A Phase 1/2 Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of ARQ 531 in Selected Subjects With Relapsed or Refractory Hematologic Malignancies
Brief Title: A Study of Nemtabrutinib (MK-1026) in Participants With Relapsed or Refractory Hematologic Malignancies (ARQ 531-101/MK-1026-001)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1026-001; ARQ 531-101 (Other: ArQule Protocol Number); MK-1026-001 (Other: MSD)
Record Dates: First submitted 2017-05-15; First posted 2017-05-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma, B-Cell; Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia; Waldenstrom Macroglobulinemia; Mantle Cell Lymphoma; Diffuse Large B Cell Lymphoma; Richter's Transformation; Follicular Lymphoma; Marginal Zone Lymphoma
Keywords: nemtabrutinib; Hematologic Malignancies; SLL; CLL; B-cell NHL; WM; BTK (Brutons tyrosine kinase); cancer; refractory; relapsed; Acalabrutinib; ArQule; BGB-3111; Blood Protein Disorders; Follicular Lymphoma; BTK Intolerant; C481; C481S; C481S Mutation; Cardiovascular Diseases; Chronic Lymphocytic Leukemia; DLBCL (Diffuse Large B-cell lymphoma); GS-4059; Hemorrhagic Disorders; Hemostatic Disorders; Ibrutinib; Immune System Diseases; Immunoproliferative Disorders; Leukemia; Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Lymphoid; Lymphatic Diseases; Lymphoma; Lymphoma, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Mantle Cell Lymphoma; Marginal zone lymphoma; Neoplasms; Neoplasms by Histologic Type; Neoplasms, Plasma Cell; NHL (Non-Hodgkins Lymphoma); ONO-4059; Paraproteinemias; Small Lymphocytic Lymphoma; Tirabrutinib; Vascular Diseases; Waldenstrom Macroglobulinemia; Zanubrutinib
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Hematologic Neoplasms; Neoplasms; Recurrence; Blood Protein Disorders; Cardiovascular Diseases; Dendritic Cell Sarcoma, Interdigitating; Hemorrhagic Disorders; Hemostatic Disorders; Immune System Diseases; Immunoproliferative Disorders; Leukemia; Leukemia, B-Cell; Leukemia, Lymphoid; Lymphatic Diseases; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Neoplasms by Histologic Type; Neoplasms, Plasma Cell; Paraproteinemias; Vascular Diseases | interventions — ARQ531

STUDY DESIGN:
Intervention Model Description: Single group assignment (definition : A type of intervention model describing a clinical trial in which all participants receive the same intervention/treatment.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Phase 1: Dose Escalation and Determination of RP2D (Experimental): Phase I: Dose Escalation and determination of RP2D, multiple dose levels of nemtabrutinib to be evaluated (Up to approximately 22 months).
  Interventions: Drug: Nemtabrutinib
- Phase 2: Expansion Cohort A (Experimental): Relapsed/Refractory chronic lymphocytic leukemia/small lymphocytic lymphoma (R/R CLL/SLL) participants with at least 2 prior systemic therapies and previously treated with a covalent Bruton's tyrosine kinase inhibitor (BTKi) who must have a documented BTK mutation on C481 residue receive up to 65 mg of nemtabrutinib per day orally in each cycle (Cycle length = 28 days) until progressive disease (PD), unacceptable adverse events (AEs), or discontinuation at investigator's discretion (up to approximately 64 months).
  Interventions: Drug: Nemtabrutinib
- Phase 2: Expansion Cohort B (Experimental): R/R CLL/SLL participants who have failed or were intolerant to a BTKi with documentation of the absence of BTK mutation on C481 residue receive up to 65 mg of nemtabrutinib per day orally in each cycle (Cycle length = 28 days) until PD, unacceptable AEs, or discontinuation at investigator's discretion (up to approximately 64 months).
  Interventions: Drug: Nemtabrutinib
- Phase 2: Expansion Cohort C (Experimental): Richter's transformation (RT) participants who have failed at least one prior therapy receive up to 65 mg of nemtabrutinib per day orally in each cycle (Cycle length = 28 days) until PD, unacceptable AEs, or discontinuation at investigator's discretion (up to approximately 64 months).
  Interventions: Drug: Nemtabrutinib
- Phase 2: Expansion Cohort D (Experimental): Follicular Lymphoma (FL) participants who have failed at least 2 prior systemic therapies and are histology grade 1, 2, or 3A receive up to 65 mg of nemtabrutinib per day orally in each cycle (Cycle length = 28 days) until PD, unacceptable AEs, or discontinuation at investigator's discretion (up to approximately 64 months).
  Interventions: Drug: Nemtabrutinib
- Phase 2: Expansion Cohort E (Experimental): Mantle Cell Lymphoma (MCL) participants who have failed at least 2 prior systemic therapies receive up to 65 mg of nemtabrutinib per day orally in each cycle (Cycle length = 28 days) until PD, unacceptable AEs, or discontinuation at investigator's discretion (up to approximately 64 months).
  Interventions: Drug: Nemtabrutinib
- Phase 2: Expansion Cohort F (Experimental): Marginal Zone Lymphoma (MZL) participants who have failed at least 2 prior systemic therapies receive up to 65 mg of nemtabrutinib per day orally in each cycle (Cycle length = 28 days) until PD, unacceptable AEs, or discontinuation at investigator's discretion (up to approximately 64 months).
  Interventions: Drug: Nemtabrutinib
- Phase 2: Expansion Cohort G (Experimental): High-grade B-cell lymphoma (BCL) participants who have failed at least 2 prior systemic therapies and have known MYC and BCL2 and/or BCL6 translocations confirmed by flourescence in situ hybridization (FISH) or overexpression by immunohistochemistry (IHC) receive up to 65 mg of nemtabrutinib per day orally in each cycle (Cycle length = 28 days) until PD, unacceptable AEs, or discontinuation at investigator's discretion (up to approximately 64 months).
  Interventions: Drug: Nemtabrutinib
- Phase 2: Expansion Cohort H (Experimental): Waldenström macroglobulinemia (WM) participants who have failed at least 2 prior systemic therapies receive up to 65 mg of nemtabrutinib per day orally in each cycle (Cycle length = 28 days) until PD, unacceptable AEs, or discontinuation at investigator's discretion (up to approximately 64 months).
  Interventions: Drug: Nemtabrutinib
- Phase 2: Expansion Food Effect Cohort I (Experimental): B-cell Non-Hodgkin's lymphoma (NHL), CLL/SLL and WM participants receive up to 65 mg of nemtabrutinib fasted (1 hour prior to or 2 hours after meal) and non-fasted per day orally in each cycle (Cycle length = 28 days) until PD, unacceptable AEs, or discontinuation at investigator's discretion (up to approximately 64 months).
  Interventions: Drug: Nemtabrutinib

INTERVENTIONS:
Drug: Nemtabrutinib — Nemtabrutinib will be orally administered once per day under fasted conditions (1 hour prior to or 2 hours after a meal) and is available in tablets in strengths of 5 mg or 20 mg. For Expansion Food Effect Cohort I, nemtabrutinib will be orally administered once per day under fasted and non-fasted condition.
  Other Names: ARQ 531; MK-1026

SUMMARY:
This study aims to evaluate the safety, tolerability, pharmacodynamic, and pharmacokinetic (PK) of nemtabrutinib (formerly ARQ 531) tablets in selected participants with relapsed or refractory hematologic malignancies. No formal hypothesis testing will be performed for this study.

DETAILED DESCRIPTION:
This study includes 2 parts: Phase 1 (dose escalation) and Phase 2 (dose expansion). In Phase 1, participants will enroll using 3+3 dose escalation design. The starting dose of nemtabrutinib in oral tablet form was 5mg/day continuously. Dose escalation will continue until the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) and dosing schedule is reached based on protocol-defined dose limiting toxicity (DLT). After the determination of the RP2D, 9 expansion cohorts will be initiated to evaluate the safety, tolerability, and efficacy of nemtabrutinib at RP2D in participants with specifically defined disease.

ELIGIBILITY:
Inclusion Criteria

Each prospective participant must meet ALL of the following inclusion criteria in order to be eligible for this study:

* Signed written informed consent granted prior to initiation of any study-specific procedures
* For the dose escalation cohorts, relapsed or refractory (R/R) participants with a diagnosis of B-cell Non-Hodgkin's lymphoma (NHL), chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL) and Waldenstrom macroglobulinemia (WM) who have received at least two prior systemic therapies . Participants must have failed or are intolerant to standard therapies and cannot be a candidate for standard salvage regimens. Participants with low grade lymphoma must be progressing and requiring treatment
* For the expansion cohorts, the following criteria must be met:

  * Cohort A: R/R CLL/SLL participants with at least 2 prior systemic therapies and previously treated with a covalent Bruton's tyrosine kinase inhibitor (BTKi) who must have a documented Bruton's tyrosine kinase (BTK) mutation on C481 residue
  * Cohort B: R/R CLL/SLL participants who have failed or were intolerant to a BTKi with documentation of the absence of BTK mutation on C481 residue. In this study, intolerance to standard therapy is defined as having experienced a grade 3 or higher adverse event that was caused by the standard therapy and resulted in treatment discontinuation
  * Cohort C: Richter's transformation (RT) participants who have failed at least one prior therapy
  * Cohort D: Follicular Lymphoma (FL) participants who have failed at least 2 prior systemic therapies and are histology grade 1, 2, or 3A
  * Cohort E: Mantle Cell Lymphoma (MCL) participants who have failed at least 2 prior systemic therapies
  * Cohort F: Marginal Zone Lymphoma (MZL) participants who have failed at least 2 prior systemic therapies
  * Cohort G: High-grade B-cell lymphoma participants who have failed at least 2 prior systemic therapies and have known MYC and BCL2 and/or BCL6 translocations
  * Cohort H: WM participants who have failed at least 2 prior systemic therapies
  * Cohort I (Food Effect): relapsed or refractory participants with a diagnosis of B-cell NHL, CLL/SLL or WM who have received at least 2 prior systemic therapies, or 1 prior therapy for RT participants. Participants must have failed or are intolerant to standard therapies and cannot be a candidate for standard salvage regimens. Participants with low grade lymphoma must be progressing and requiring treatment.
* Disease status requirement:

  * For CLL participanst symptomatic disease that mandates treatment (Hallek et al. 2018)
  * For B-cell NHL participants, measurable disease by imaging scan
  * For WM, serum immunoglobulin M (IgM) with a minimum IgM level of ≥ 2 times the upper limit of normal (ULN)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Good organ function
* Creatinine clearance of ≥ 60 mL/min as estimated by the Cockcroft-Gault equation or by 24-hour urine collection
* Total bilirubin ≤ 1.5 x institutional ULN (total bilirubin of ≤ 3 x institutional ULN in participants with documented Gilbert's syndrome)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × institutional ULN
* Platelet count ≥ 50,000/µL
* Absolute neutrophil count (ANC) ≥ 1000/µL
* Hemoglobin (Hgb) ≥ 8.0 g/dL, stable for ≥ 1 week.
* For men and women of child-bearing potential, willing to use adequate contraception (e.g., latex condom, cervical cap, diaphragm, abstinence, etc.) for the entire duration of the study
* Female participants of child-bearing potential must have a negative serum pregnancy test within 14 days of the first day of drug dosing
* Ability to swallow oral medications without difficulty

Exclusion Criteria

Potential participants who meet ANY of the following exclusion criteria are not eligible for enrollment into this study:

* Had immunotherapy, radiotherapy, radioimmunotherapy, biological therapy, chemotherapy, or treatment with an investigational product within 5 half-lives or four weeks (whichever is shorter) prior to treatment initiation, or oral therapy within 5 half-lives or one week (whichever is shorter) prior to treatment initiation
* Transformation of follicular lymphoma (FL) to a more aggressive subtype of lymphoma or grade 3b FL
* Participants currently being treated with the following drugs:

  * CYP2C8 substrates with a narrow therapeutic index (such as paclitaxel)
  * P-gp substrates with a narrow therapeutic index (such as digoxin)
  * CYP3A strong inducers (such as rifampin) Note: A washout period of at least 5 times the half-life after the last dose of any of the above treatments is required for a participant to be eligible for study enrollment
* Active central nervous system (CNS) involvement
* Pregnant or breast-feeding women
* Has significant, ongoing co-morbid conditions which would preclude safe delivery of the study drug
* Uncontrolled illness including but not limited to ongoing or active infection, symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or IV heart failure), unstable angina pectoris, cardiac arrhythmia, cardiac infarction in the past six months, and psychiatric illness that would limit compliance with study requirements
* QT corrected (QTc) prolongation (defined as a QTc > 450 msecs) or other significant electrocardiogram (ECG) abnormalities including 2nd degree atrioventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min).
* Active Hepatitis B or Hepatitis C infection.
* Other medical or psychiatric illness or organ dysfunction which, in the opinion of the Investigator, would either compromise the participant's safety or interfere with the evaluation of the safety of the study agent
* History of prior cancer within < 1 year, except for basal cell or squamous cell carcinoma of the skin, cervical cancer in situ or other in situ carcinomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants Experiencing Dose Limiting Toxicity (DLT) | Cycle 1 (up to 28 days)
  DLT is defined by the occurrence of any of the following treatment emergent adverse event (TEAE) unless unequivocally due to the underlying malignancy or an extraneous cause within the first 28 days of study treatment (for dose escalation only) and graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. Any Grade 5 TEAE, any Grade 3 nonhematological TEAE except alopecia, nausea, vomiting, diarrhea, and transient Grade 3 laboratory abnormalities which recover within 1 week without intervention, any Grade 3 hematological TEAE that does not recover to Grade 1 or baseline within 7 days with the exception of Grade 3 lymphocytosis, which is considered to be an expected outcome of BTK inhibition, any Grade 4 nonhematological and hematological TEAE, or any other toxicity that in the view of the investigator represents a clinically significant hazard to the participant.
Phase 1: Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 86 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE will be reported.
Phase 1: Number of Participants Who Discontinued Study Treatment Due to an AE | Up to approximately 86 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE will be reported.
Phase 2: Expansion Cohorts A, B & C: Objective Response Rate (ORR) per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Criteria as Assessed by the Investigator | Up to approximately 64 months
  ORR is defined as the percentage of participants achieving a best overall response of complete response (CR), partial response (PR) or partial response with lymphocytosis (PRL). iwCLL criteria as assessed by the investigator. CR is defined as meeting the following criteria: no lymph nodes >1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or ≥50% increase from screening, hemoglobin >11 g/dL or ≥50% increase from screening, CLL cells or B lymphoid nodules in marrow.
Phase 2: Expansion Cohorts A, B, C: ORR per Lugano Classification as Assessed by the Investigator | Up to approximately 64 months
  ORR is defined as percentage of participants achieving best overall response of CR/PR per Lugano classification as assessed by investigator. CR defined as EITHER CR by imaging (computed tomography [CT]): all lymph nodes normal (none ≥15 mm) & normal liver, spleen OR complete metabolic response (CMR): score of 1, 2 or3 on 5-point scale assessing fluorodeoxyglucose (FDG) metabolic activity in lymphomatous lesions (range: 1=no uptake above background to 5=uptake markedly higher than liver) AND bone marrow (BM) normal by morphology. PR defined as EITHER PR by imaging (CT) with ≥50% decrease in sum of product of diameters [SPD] of target lesions, no worsening of nontarget lesions, no new lesions and ≥50% spleen abnormal portion OR Partial Metabolic Response (PMR) with score of 4/5 on FDG 5-point scale (with no new lesions) & decreased overall uptake AND residual BM abnormalities; OR CR by imaging with residual BM abnormalities; OR PR by imaging without residual BM abnormalities.

SECONDARY OUTCOMES:
Phase 2: Number of Participants Who Experienced an AE | Up to approximately 64 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE will be reported.
Phase 2: Number of Participants Who Discontinued Study Treatment Due to an AE | Up to approximately 64 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE will be reported.
Time to Maximum Concentration (Tmax) of Nemtabrutinib | Cycles 1-92: Days 1, 2: Predose and up to 16 hours postdose (each cycle length = 28 days, up to approximately 86 months)
  Blood samples will be collected at prespecified time points to determine Tmax of nemtabrutinib.
Maximum Concentration (Cmax) of Nemtabrutinib | Cycles 1-92: Days 1, 2: Predose and up to 16 hours postdose (each cycle length = 28 days, up to approximately 86 months)
  Blood samples will be collected at prespecified time points to determine Cmax of nemtabrutinib.
Area Under the Concentration-Time Curve From Time Zero to 24 Hours (AUC 0-24hrs)of Nemtabrutinib | Cycles 1-92: Days 1, 2: Predose and up to 24 hours postdose (each cycle length = 28 days, up to approximately 86 months)
  Blood samples will be collected at prespecified time points to determine AUC 0-24hrs of nemtabrutinib.
Terminal Elimination Half-Life (t1/2) of Nemtabrutinib | Cycles 1-92: Days 1, 2: Predose and up to 16 hours postdose (each cycle length = 28 days, up to approximately 86 months)
  t1/2 is the time it takes for the concentration of nemtabrutinib in the body to decrease by half during the elimination phase.
Phase 2: Expansion Cohorts D-H: ORR per iwCLL Criteria as Assessed by the Investigator | Up to approximately 64 months
  ORR is defined as the percentage of participants achieving a best overall response of complete response (CR), partial response (PR) or partial response with lymphocytosis (PRL). iwCLL criteria as assessed by the investigator. CR is defined as meeting the following criteria: no lymph nodes >1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or ≥50% increase from screening, hemoglobin >11 g/dL or ≥50% increase from screening, CLL cells or B lymphoid nodules in marrow.
Phase 2: Expansion Cohorts D-H: ORR per Lugano classification as Assessed by the Investigator | Up to approximately 64 months
  ORR is defined as percentage of participants achieving best overall response of CR/PR per Lugano classification as assessed by investigator. CR defined as EITHER CR by imaging (computed tomography [CT]): all lymph nodes normal (none ≥15 mm) & normal liver, spleen OR complete metabolic response (CMR): score of 1, 2 or3 on 5-point scale assessing fluorodeoxyglucose (FDG) metabolic activity in lymphomatous lesions (range: 1=no uptake above background to 5=uptake markedly higher than liver) AND bone marrow (BM) normal by morphology. PR defined as EITHER PR by imaging (CT) with ≥50% decrease in sum of product of diameters [SPD] of target lesions, no worsening of nontarget lesions, no new lesions and ≥50% spleen abnormal portion OR Partial Metabolic Response (PMR) with score of 4/5 on FDG 5-point scale (with no new lesions) & decreased overall uptake AND residual BM abnormalities; OR CR by imaging with residual BM abnormalities; OR PR by imaging without residual BM abnormalities.
Phase 2: Expansion Cohorts A, B, H: Duration of Response (DOR) per iwCLL Criteria as Assessed by the Investigator | Up to approximately 64 months
  DOR is defined as the time from the first documented evidence of CR or PR (or PRL for CLL/SLL participants) until progressive disease or death due to any cause, whichever occurs first. CR is defined as meeting the following criteria: no lymph nodes >1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or ≥50% increase from screening, hemoglobin >11 g/dL or ≥50% increase from screening, CLL cells or B lymphoid nodules in marrow.
Phase 2: Expansion Cohorts C-G: DOR per Laguna Classification As Assessed by Investiigator | Up to approximately 64 months
  DOR is defined as time from first documented evidence of CR/PR (or PRL for CLL/SLL participants) until progressive disease or death due to any cause, whichever occurs first. CR defined as EITHER CR by imaging (computed tomography [CT]): all lymph nodes normal (none ≥15 mm) & normal liver, spleen OR complete metabolic response (CMR): score of 1, 2 or3 on 5-point scale assessing FDG metabolic activity in lymphomatous lesions (range: 1=no uptake above background to 5=uptake markedly higher than liver) AND BM normal by morphology. PR defined as EITHER PR by imaging (CT) with ≥50% decrease in SPD of target lesions, no worsening of nontarget lesions, no new lesions and ≥50% spleen abnormal portion OR PMR with score of 4/5 on FDG 5-point scale (with no new lesions) & decreased overall uptake AND residual BM abnormalities; OR CR by imaging with residual BM abnormalities; OR PR by imaging without residual BM abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (10):
- United States (10):
  - Mayo Clinic Hospital ( Site 0140), Scottsdale, Arizona
  - UCLA Hematology & Oncology ( Site 0017), Los Angeles, California
  - Colorado Blood Cancer Institute ( Site 0225), Denver, Colorado
  - University of Michigan ( Site 0018), Ann Arbor, Michigan
  - Mayo Clinic - Rochester ( Site 0138), Rochester, Minnesota
  - Duke Cancer Center ( Site 0067), Durham, North Carolina
  - The Ohio State University Wexner Medical Center ( Site 0056), Columbus, Ohio
  - Tennessee Oncology, PLLC ( Site 0020), Nashville, Tennessee
  - UT Southwestern Medical Center ( Site 0116), Dallas, Texas
  - University of Utah, Huntsman Cancer Institute ( Site 0122), Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Woyach JA, Stephens DM, Flinn IW, Bhat SA, Savage RE, Chai F, Eathiraj S, Reiff SD, Muhowski EM, Granlund L, Szuszkiewicz L, Wang W, Schwartz B, Ghori R, Farooqui MZH, Byrd JC. First-in-Human Study of the Reversible BTK Inhibitor Nemtabrutinib in Patients with Relapsed/Refractory Chronic Lymphocytic Leukemia and B-Cell Non-Hodgkin Lymphoma. Cancer Discov. 2024 Jan 12;14(1):66-75. doi: 10.1158/2159-8290.CD-23-0670. PMID 37930156
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/